CLINICAL TRIAL: NCT01567267
Title: Phase II Study of a Short Term Educational Intervention for Upcoming Biology Teachers to Teach Principles of Evidence-based Medicine (EbM) in Biology Classes at High-school
Brief Title: Evaluation of Educational Intervention to Teach Principles of Evidence-based Medicine (EbM) in Biology Classes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Reinhard Strametz, MD, EbM Working Group, Institute for General Practice, Faculty of Medicine, Goethe University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EbM@Bio-01
Record Dates: First submitted 2012-03-14; First posted 2012-03-30 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: Evidence-based Medicine; Good Scientific Practice; Problem-based Learning; Critical health literacy; Educational intervention
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental educational intervention (Experimental): Experimental educational intervention
  Interventions: Behavioral: Experimental educational intervention
- Standard educational intervention (Active Comparator): Standard educational intervention
  Interventions: Behavioral: Standard educational intervention

INTERVENTIONS:
Behavioral: Experimental educational intervention — Educational intervention consisting of a 4-day-course in Evidence-based Medicine and Good Scientific Practice combined with the method of Problem-based Learning.
  Arms: Experimental educational intervention
Behavioral: Standard educational intervention — Educational intervention on the didactics of biology (4-day-course) not containing elements of Evidence-based Medicine, Good Scientific Practice or Problem-based learning.
  Arms: Standard educational intervention

SUMMARY:
The purpose of this study is to identify the effect of a short term educational intervention for upcoming biology teachers to teach principles of Evidence-based Medicine (EbM) and Good Scientific Practice (GSP) to high-school biology students.

DETAILED DESCRIPTION:
Shared decision making is increasingly demanded by patients in order to take part in health care decisions. However this demand for autonomy can only be used for shared decision making if the patient has basic skills in critical health literacy. To transfer health care literacy to young and healthy consumers educational intervention programs at high-school might be a feasible and effective way. This preliminary phase 2 study is designed to investigate the effect of an educational intervention to be integrated in a curriculum for upcoming teachers in biology.

ELIGIBILITY:
Inclusion Criteria:

* students becoming biology teachers at participating university during enrollment period

Exclusion Criteria:

* refusal to participate in study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2010-02; Primary Completion 2018-09 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Difference in knowledge about EbM/GSP | Before (day1), during (day 2) and after (day 4) intervention
  Difference in knowledge about EbM/GSP measured by alternating standardized, pre-validated, single-best/short-answer questionnaires consisting of 20 questions each

SECONDARY OUTCOMES:
Difference in skills about critically appraising scientific literature | Before (day 1), during (day 2) and after (day 4) intervention
  Difference in skills about critically appraising scientific literature measured by alternating randomized-controlled trials evaluated by a standardized checklist related to items of the CONSORT statement.
Skills in teaching principles of EbM and GSP to high school students in intervention group | After educational intervention (day 5)
  Skill in teaching principles of EbM and GSP are evaluated for preparation of lessons using a standardized preparation form and performance of lessons evaluated by transcription of video tapes from each participant in the intervention group using a consented evaluation catalogue
Overall acceptance of educational intervention study participants | During (day 2) and after intervention (day 4)
  Overall acceptance of educational intervention is evaluated by standardized questionnaires at day 2 and day 4 in the educational intervention group.
Overall acceptance of study lessons for biology high-school students | After study lessons (day 5)
  Overall acceptance of study lessons for biology high-school students is evaluated by a standardized questionnaire at day 5.

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Strametz, MD, Principal Investigator — EbM Working Group, Institute for General Practice, Faculty of Medicine, Goethe University, Frankfurt/Germany
Locations (1):
- University of Siegen, Section of biology and und their didactics, Siegen, Germany

REFERENCES:
- [Derived] Matic-Strametz M, Strametz R, Bohrt K, Ochsendorf F, Weberschock T. [Students in Training to Become Biology Teachers - a controlled phase II trial (NCT01567267)]. Z Evid Fortbild Qual Gesundhwes. 2013;107(1):53-61. doi: 10.1016/j.zefq.2012.11.017. Epub 2012 Dec 7. German. PMID 23415344